CLINICAL TRIAL: NCT01565577
Title: Phase 3, Vaccinal Activity Assessment of MenBVac Against Nesseiria Menigitidis B:14,P1.7,16 Strain in Child Vaccinated With MenBVac®
Brief Title: Evaluation of Immune Response Against the Strain of Neisseria Meningitidis B: 14, P1-7, 16 Patients Vaccinated With MenBVac® (Extension MenbVac)
Acronym: Exten MenbVac
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Direction Générale de la Santé, France (Other); Institut Pasteur (Industry); Dieppe (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2011/199/HP
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Vaccination With MenbVac
Keywords: Neisseria meningitidis B:14, P1-7, 16; Serum bactericidal activity; Menbvac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bras A (Experimental)
  Interventions: Biological: MenbVac

INTERVENTIONS:
Biological: MenbVac — Blood test

SUMMARY:
This study aims to estimate the vaccinal immunity four years after four doses of MenbVac in children aged 4-8 years.

ELIGIBILITY:
Inclusion Criteria:

* children born between 01/01/2000 and 06/23/2005, living in Dieppe-Est, Dieppe-Ouest and Offranville, vaccinated with four doses of MenBVac in the first MenbVac clinical trial study,
* parental authority(ies)assent.

Exclusion Criteria:

* no parental authority(ies)assent,
* no parental authority(ies)assent,
* no blood sample during the third vaccination,
* impossibility of third vaccination.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
vaccine Immunity | two and a half years after the fouth vaccination
  assessment of vaccine Immunity with measure of percentage of children with an hSBA title >= 4 four years after four doses of MenbVac

CONTACTS AND LOCATIONS:
Overall Officials: François Caron, Professor, Principal Investigator — CHU - Hôpitaux de Rouen
Locations (1):
- UH-rouen, Rouen, Seine Maritime, France